CLINICAL TRIAL: NCT02315625
Title: A Phase II Trial of Mutation-Targeted Therapy With Sunitinib or Everolimus in Patients With Advanced Low-or Intermediate Grade Neuroendocrine Tumors of the Gastrointestinal Tract and Pancreas With or Without Cytoreductive Surgery
Brief Title: Study of Mutation-Targeted Therapy With Sunitinib or Everolimus in People With Advanced Low- or Intermediate-Grade Neuroendocrine Tumors of the Gastrointestinal Tract and Pancreas With or Without Cytoreductive Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study closed due to poor accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Naris Nilubol, M.D., National Cancer Institute, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 150040; 15-C-0040
Record Dates: First submitted 2014-12-11; First posted 2014-12-12 (Estimated); Results first posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: Neuroendocrine Tumors; Neuroendocrine Carcinoma; Neuroendocrine Neoplasms; Carcinoma, Neuroendocrine; Neuroendocrine Tumors of the Gastrointestinal Tract and Pancreas
Keywords: MEN1; VHL; Neoplasm; NF1; mTOR
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoma, Neuroendocrine; Neoplasms | interventions — Sunitinib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/ Arm 1 Sunitinib (Experimental): Sunitinib
  Interventions: Drug: Sunitinib
- 2/ Arm 2 Everolimus (Experimental): Everolimus
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Sunitinib — 37.5 mg once daily will continue until progression or unacceptable treatment-related toxicity
  Other Names: SU11248
  Arms: 1/ Arm 1 Sunitinib
Drug: Everolimus — 10 mg daily will continue until progression or unacceptable treatment-related toxicity
  Other Names: Afinitor
  Arms: 2/ Arm 2 Everolimus

SUMMARY:
Background:

- Neuroendocrine tumors (NETs) come from cells of the hormonal and nervous systems. Some people have surgery to shrink the tumor. Sometimes the tumors come back. Researchers think that treatment with drugs based on knowing the defective gene might give better results.

Objective:

- To see if drugs selected based on the defective gene result in better tumor response. The drugs are Sunitinib and Everolimus.

Eligibility:

- People age 18 and older with an advanced low- or intermediate-grade gastrointestinal or pancreatic neuroendocrine tumor.

Design:

* Participants will be screened with:
* Medical history
* Physical exam
* Scans
* Blood, urine, and lab tests
* The study team will see if participants should have surgery.
* If yes, participants will:
* Sign a separate consent
* Have computed tomography (CT) scan before and after surgery
* Have as much of the tumor removed as possible. A small piece will be tested for mutation type.
* If no, participants will have a small piece of tumor removed for the testing.
* If the surgery might cure them, the participant will leave the study. The other participants will be assigned to take either Sunitinib or Everolimus.
* Participants will take their drug by mouth once a day. They will keep a medicine diary. Some will keep track of their blood pressure at least weekly.
* Screening tests may be repeated at study visits. Participants also may have their heart evaluated.
* About 30 days after the last day of their study drug, participants will have a follow-up visit that repeats the screening tests.
* Participants will be contacted every 3 months after this visit.

DETAILED DESCRIPTION:
Background:

* Neuroendocrine tumors (NETs) of the gastrointestinal tract and pancreas are a rare and heterogeneous group of neoplasms with unique tumor biology, natural history, and clinical management issues.
* Most NETs are sporadic, but they can be part of familial cancer syndromes such as multiple endocrine neoplasia type 1 (MEN1), neurofibromatosis type 1 (NF1) or Von Hippel-Lindau (VHL) syndrome.
* Well-differentiated, low or intermediate grade NETs have a heterogeneous natural history.
* Surgery is the only curative treatment option in patients with localized early stage NETs.
* The optimal management strategy for patients with advanced NETs is unknown.
* The majority of NETs have somatic mutations in MEN1 and cyclin dependent kinase inhibitor 1B (CDKN1B), and genes involved in the phosphatidylinositol-3-kinase (PI3K/AKT/mammalian target of rapamycin (mTOR) signaling pathway, and/or overexpression of growth factors and their receptors such as vascular endothelial growth factor (VEGF), vascular endothelial growth factor receptors (VEGFR), platelet-derived growth factor (PDGF), and platelet-derived growth factor receptors (PDGFR) that can be targeted for therapy.
* Survival in patients with NETs and somatic mutations is better than patients with wild type NETs.
* Sunitinib (multi-tyrosine kinase inhibitor) and Everolimus (mTOR signaling pathway inhibitor) are currently approved for the treatment of progressive, unresectable, locally advanced or metastatic pancreatic NETs.
* However, mutation targeted therapy with Sunitinib or Everolimus has not been studied in this patient population.
* The present proposal aims to determine if mutation targeting therapy for patients with advanced low- or intermediate grade NETs is more effective than historically expected results.

Objectives:

-To determine the progression-free survival in patients with NETs of the gastrointestinal tract and pancreas treated with Sunitinib or Everolimus based on tumor genotyping.

Eligibility:

-Patients with:

* progressive, histologically or cytologically diagnosed low or intermediate grade locally advanced or metastatic NETs.
* Age greater than or equal to 18 years

Design:

* Phase II open labeled clinical trial.
* Tumor biopsy for tumor genotyping will be performed if the patient does not have archival tissue available and does not have MEN1, VHL or NF1.
* Patients with somatic or germline mutations in MEN1/PDGFR/KIT/FMS-like tyrosine kinase-3 will be treated with Sunitinib. (Arm 1)
* Patients with somatic/germline mutations in NF1/PTEN/PI3K/AKT/mTOR/VHL will be treated with Everolimus. (Arm 2)
* Patients with wildtype tumor will be treated with Sunitinib. (Arm 1)
* Patients who have disease-progression on either Sunitinib or Everolimus will cross-over to the other drug.
* Treatment will continue until disease progression, unacceptable toxicity, or consent withdrawal.
* Up to 120 patients will be accrued to the study. It is anticipated that 20-30 patients per year may enroll into this trial; thus accrual may be completed in 4-5 years.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Progressive, histologically or cytologically diagnosed low or intermediate grade, neuroendocrine tumors confirmed by the Laboratory of Pathology, National Cancer Institute (NCI). Disease progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria for progression of disease or any new lesions seen on 68-Gallium DOTATATE within the 18 months prior to enrolment.
2. Age greater than or equal 18 years, because the incidence and prevalence of metastatic pancreatic and gastrointestinal neuroendocrine tumors in the pediatric patient population is exceedingly rare (children are excluded from this study, but will be eligible for future pediatric trials).
3. Patients must have measurable disease according to RECIST criteria on anatomic imaging studies (computed tomography (CT) scan or magnetic resonance imaging (MRI)).
4. Willingness to undergo tumor biopsy if the patient does not have a known familial cancer syndrome (multiple endocrine neoplasia type 1 (MEN1), Von Hippel-Lindau (VHL) and neurofibromatosis type 1 (NF1)). Archival tissue available.
5. Eastern Cooperative Oncology Group (ECOG) performance status <2.
6. Patients must have normal organ and bone marrow function as defined below:

   * hemoglobin greater than or equal 9 g/dL *
   * leukocytes greater than or equal 3,000/mcL *
   * absolute neutrophil count greater than or equal 1,500/mcL *
   * platelets greater than or equal institutional lower limit of normal
   * total bilirubin within normal institutional limits
   * Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamic-pyruvic transaminase (SGPT) less than or equal 2.5 times institutional upper limit of normal

   (less than or equal 5 times upper limit of normal (ULN) in patients with liver metastases)

   - creatinine within normal institutional limits

   OR
   * creatinine clearance greater than or equal 60 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal.
   * International Normalized Ratio (INR) less than or equal 2;

     * If a patient's bone marrow function falls below the indicated values and it is not thought to be related to prior treatments a hematology consult will be ordered. If Hematology deems the patients safe to proceed with treatment they will be allowed to enroll on study. In such cases, the patients absolute neutrophil count must be greater than 1,000/mcl, hemoglobin must be greater than 7.5 g/dL and the platelet count must be > 75,000 mcL. Each patient will also be seen by a medical oncologist at follow-up visits if possible.
7. Fasting serum cholesterol less than or equal 300 mg/dL OR less than or equal 7.75 mmol/L AND fasting triglycerides less than or equal 2.5x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication;
8. Women of childbearing potential (WOCBP) or partners of WOCBP participating in this study must agree to use highly effective contraception while on treatment and for at least 8 weeks after end of treatment, because the effects of Sunitinib and Everolimus on the developing human fetus are unknown. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

   Highly effective contraception methods include combination of:
   1. Any two of the following:

      * Use of oral, injected or implanted hormonal methods of contraception or;
      * Placement of an intrauterine device (IUD) or intrauterine system (IUS);
      * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository;
   2. Total abstinence or;
   3. Male/female sterilization.

   Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to enrollment. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential.
9. Must have fully recovered from toxicities of any prior treatment with cytotoxic drugs, radiotherapy, surgery, or other anti-cancer modalities (returned to baseline status as noted before most recent treatment or less than or equal grade 1).
10. Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Uncontrolled hypertension (>150/100 mmHg).
* Prior external beam radiation therapy to the target lesion(s) within 1 months prior to enrollment
* Prior systemic chemotherapy or therapy with one of the investigational agents within 1 month prior to enrollment.
* Patients who had therapy with one of the investigational agents more than 1 month prior to enrollment in whom tumor genotyping show assignment to the same investigational agent.
* Patients who are receiving any other investigational agents.
* Patients with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Sunitinib or Everolimus.
* Patients who have any severe and/or uncontrolled medical conditions such as:

  1. unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction less than or equal 6 months prior to start of Everolimus, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease
  2. symptomatic congestive heart failure of New York heart Association Class III or IV
  3. active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease
  4. known severely impaired lung function
  5. Corrected QT interval (QTc) interval > 450 msec for males or > 470 msec for females
  6. active, bleeding diathesis;
  7. psychiatric illness/social situations that would preclude informed consent, limit compliance with study requirements
* Pregnant or nursing patients will be excluded from the study, because the effects of Sunitinib and Everolimus on the developing human fetus are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Sunitinib or Everolimus, breastfeeding should be discontinued if the mother is treated with Sunitinib or Everolimus.
* Current treatment with therapeutic doses of Coumadin-derivative anticoagulants (low dose Coumadin up to 2 mg by mouth (PO) daily for deep vein thrombosis prophylaxis is allowed).
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with study agents.
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome, or the inability to take oral medication
* Uncontrolled diabetes mellitus as defined by hemoglobin A1C (HbA1c) >8% despite adequate therapy. Patients with a known history or diagnosis of diabetes mellitus who are on therapy and have had good blood sugar control may be included, even if the HbA1c is > 8% because this value can take up to 3-4 months to normalize
* Patients who have received live attenuated vaccines within 1 week of start of Everolimus and during the study. Patient should also avoid close contact with others who have received live attenuated vaccines. Examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, Bacille Calmette-Guerin (BCG), yellow fever, varicella and TY21a typhoid vaccines
* Patients who are on chronic treatment with corticosteroids or other immunosuppressive agents (topical or inhaled corticosteroids are allowed)
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study
* Patients who are taking medications that are strong inhibitors of cytochrome P450 AA4 (CYP3A4) or PgP and need to remain on these medications. For a current table of Substrates, Inhibitors and Inducers please access the following website:http://www.fda.gov/Drugs/DevelopmentApprovalProcess/DevelopmentResourc es/DrugInteractionsLabeling/ucm093664.htm
* Patients who have a history of another primary malignancy from which the patient has been disease free for < 3 years at the time of enrolment, with the exceptions of: a patient with a familial cancer syndrome-associated NETs including MEN1, VHL, NF-1, and tuberous sclerosis (TS);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-04-08 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naris Nilubol, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gan HK, Seruga B, Knox JJ. Sunitinib in solid tumors. Expert Opin Investig Drugs. 2009 Jun;18(6):821-34. doi: 10.1517/13543780902980171. PMID 19453268
- [Background] Tanaka C, O'Reilly T, Kovarik JM, Shand N, Hazell K, Judson I, Raymond E, Zumstein-Mecker S, Stephan C, Boulay A, Hattenberger M, Thomas G, Lane HA. Identifying optimal biologic doses of everolimus (RAD001) in patients with cancer based on the modeling of preclinical and clinical pharmacokinetic and pharmacodynamic data. J Clin Oncol. 2008 Apr 1;26(10):1596-602. doi: 10.1200/JCO.2007.14.1127. Epub 2008 Mar 10. PMID 18332467
- [Background] Khagi S, Saif MW. Neuroendocrine tumors: treatment updates. JOP. 2013 Jul 10;14(4):367-71. doi: 10.6092/1590-8577/1657. PMID 23846929
- [Result] Neychev V, Steinberg SM, Cottle-Delisle C, Merkel R, Nilubol N, Yao J, Meltzer P, Pacak K, Marx S, Kebebew E. Mutation-targeted therapy with sunitinib or everolimus in patients with advanced low-grade or intermediate-grade neuroendocrine tumours of the gastrointestinal tract and pancreas with or without cytoreductive surgery: protocol for a phase II clinical trial. BMJ Open. 2015 May 19;5(5):e008248. doi: 10.1136/bmjopen-2015-008248. PMID 25991462
- [Result] Tirosh A, Killian JK, Zhu YJ, Petersen D, Walling J, Mor-Cohen R, Neychev V, Stevenson H, Keutgen XM, Patel D, Nilubol N, Meltzer P, Kebebew E. ONCOGENE PANEL SEQUENCING ANALYSIS IDENTIFIES CANDIDATE ACTIONABLE GENES IN ADVANCED WELL-DIFFERENTIATED GASTROENTEROPANCREATIC NEUROENDOCRINE TUMORS. Endocr Pract. 2019 Jun;25(6):580-588. doi: 10.4158/EP-2018-0603. Epub 2019 Mar 13. PMID 30865533
- [Derived] Neychev V, Sadowski SM, Zhu J, Allgaeuer M, Kilian K, Meltzer P, Kebebew E. Neuroendocrine Tumor of the Pancreas as a Manifestation of Cowden Syndrome: A Case Report. J Clin Endocrinol Metab. 2016 Feb;101(2):353-8. doi: 10.1210/jc.2015-3684. Epub 2015 Dec 17. PMID 26678657
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-C-0040.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study closed due to poor accrual.
Groups:
- Sunitinib Followed by Everolimus: In Period 1 participants received Sunitinib 37.5 mg once daily until progression or unacceptable treatment-related toxicity. In Period 2 participants received Everolimus 10 mg daily until progression or unacceptable treatment-related toxicity.
- Everolimus Followed by Sunitinib: In Period 1 participants received Everolimus 10 mg daily until progression or unacceptable treatment-related toxicity. In Period 2 participants received Sunitinib 37.5 mg once daily until progression or unacceptable treatment-related toxicity.
Period: First Intervention
Arm/Group | Sunitinib Followed by Everolimus | Everolimus Followed by Sunitinib
Started | 14 | 2
Completed | 13 | 2
Not Completed | 1 | 0
Not completed — Disease Progression | 1 | 0
Period: Second Intervention
Arm/Group | Sunitinib Followed by Everolimus | Everolimus Followed by Sunitinib
Started | 13 | 2
Completed | 9 | 1
Not Completed | 4 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Study closure | 1 | 0
Not completed — Disease Progression | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sunitinib Followed by Everolimus | Everolimus Followed by Sunitinib | Total
Number analyzed (Participants) | 14 | 2 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 0 | 12
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.94 (8.49) | 53.41 (9.73) | 53.17 (9.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 9 | 2 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 13 | 2 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 11 | 2 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 2 | 16

OUTCOME MEASURES:

1. Primary Outcome: Median Amount of Time Subject Survives Without Disease Progression After Treatment
Description: Median amount of time subject survives without disease progression after treatment. Progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) and is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progressions.
Time Frame: Up to approximately 2 years
Population: The data in this outcome measure is reported per sequence as pre-specified in the protocol.
Measure: Median (Full Range); unit: months
Groups:
- Sunitinib First, Everolimus Second: Participants who received Sunitinib first, followed by Everolimus.
- Everolimus First, Sunitinib Second: Participants who received Everolimus first, followed by Sunitinib.
Arm/Group | Sunitinib First, Everolimus Second | Everolimus First, Sunitinib Second
Number analyzed (Participants) | 14 | 2
months | 7 [3 to 15] | 18 [0 to 18]

2. Secondary Outcome: Number of Participants With an Overall Response
Description: Overall response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) is defined as Complete Response (CR), Partial Response (PR), and Stable Disease (SD). Complete Response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Stable Disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease (PD) (e.g. appearance of one or more new lesions), taking as reference the smallest sum of diameters while on study.
Time Frame: Every 3 months until disease progression, up to 12 months
Population: The data in this outcome measure is reported per sequence as pre-specified in the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib First, Everolimus Second | Everolimus First, Sunitinib Second
Number analyzed (Participants) | 14 | 2
Participants | 1 | 0

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from treatment start date until date of death or date last known alive following therapy.
Time Frame: Up to approximately 4 years
Population: The data in this outcome measure is reported per sequence as pre-specified in the protocol.
Measure: Median (Full Range); unit: Months
Arm/Group | Sunitinib First, Everolimus Second | Everolimus First, Sunitinib Second
Number analyzed (Participants) | 14 | 2
Months | 25.5 [6 to 39] | 10.7 [0.427397 to 21]

4. Secondary Outcome: Median Survival Time (MST)
Description: MST is the amount of time a subject survives after therapy.
Time Frame: Death, an average of 12 months follow up
Population: The data in this outcome measure is reported per sequence as pre-specified in the protocol.
Measure: Median (Full Range); unit: Months
Arm/Group | Sunitinib First, Everolimus Second | Everolimus First, Sunitinib Second
Number analyzed (Participants) | 14 | 2
Months | 9.5 [0.4927 to 33] | 5.5 [0 to 11]

5. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study approximately 49 months and 9 days.
Population: One participant did not receive Sunitinib and 5 did not receive Everolimus.
Measure: Count of Participants; unit: Participants
Groups:
- Sunitinib: Participants who received Sunitinib in period 1 or 2.
- Everolimus: Participants who received Everolimus in period 1 or 2.
Arm/Group | Sunitinib | Everolimus
Number analyzed (Participants) | 15 | 11
Participants | 15 | 11

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study on up to 30 days after treatment discontinuation, approximately 49 months and 9 days.
Arm/Group | Sunitinib | Everolimus
All-Cause Mortality (participants affected / at risk) | 1/15 | 1/11
Serious Adverse Events (participants affected / at risk) | 3/15 | 2/11
Other Adverse Events (participants affected / at risk) | 14/15 | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib (N=15) | Everolimus (N=11)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (3)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Eye disorders - Other, amaurosis fugax (Eye disorders) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib (N=15) | Everolimus (N=11)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (6)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (5) | 3 (5)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (6) | 2 (2)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, GI bleed, oral lesion (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (9) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (3)
Neutrophil count decreased (Investigations) | 4 (10) | 1 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (4)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (2)
White blood cell decreased (Investigations) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/25/NCT02315625/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT02315625/ICF_001.pdf